CLINICAL TRIAL: NCT00160862
Title: A Randomised, Double-Blind, Placebo-Controlled, Crossover Study to Determine the Effect of a Single Oral Dose of SLV 317 on Substance P-Induced Venodilation in the Hand Vein of Healthy Male Volunteers
Brief Title: NK-1 Antagonism of SLV317 in Humans
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Heidelberg University (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: K071
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2005-09-12 (Estimated); Status verified 2005-09

CONDITIONS: Healthy
MeSH Terms: interventions — SLV317

INTERVENTIONS:
Drug: SLV317

SUMMARY:
The primary objective is to determine the effect of a single oral dose of 250 mg SLV 317 on substance P-induced venodilation in the hand vein of healthy male volunteers as compared to placebo.

DETAILED DESCRIPTION:
This will be a double-blind, placebo-controlled, oral single dose cross-over study. 18 healthy male volunteers will receive 250 mg SLV 317 or placebo in randomised order with a minimum wash-out period of one week between the two administrations.

Pharmacodynamic assessments will be performed up to 4.25 hours post-dose using the dorsal hand vein compliance technique. After obtaining venoconstriction via infusions of phenylephrine, substance P will be co-infused intermittently to induce venodilation. Substance P infusions will be separated by intervals of 45 minutes in order to prevent the well-known occurrence of tolerance.

Venous blood sampling for pharmacokinetic evaluation will be performed up to 24 hours post-dose.

Safety will be assessed by measuring ECG, pulse rate, blood pressure, haematology, blood chemistry, urinalysis, and by monitoring of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Male non-smoking volunteers, age: 18-45, with a body mass index (BMI) in the range from 19-26 (kg/m2), inclusive
* Good health as determined by medical history, physical examination, electrocardiogram, serum/urine biochemistry and haematology
* A lying blood pressure after resting for 5 minutes between 100 150 mmHg (systolic) and 50-90 mmHg (diastolic)
* A lying heart rate (ECG) after resting for 5 minutes between 45 and 100 beats/min.
* Able and willing to give written informed consent

Exclusion Criteria:

* Known condition causing endothelial dysfunction (e.g. diabetes, hyperlipidaemia, smoking, arterial hypertension, hyperhomocysteinaemia)
* Evidence of cardiovascular, gastrointestinal/hepatic, neurologic/psychiatric, respiratory, urogenital, haematologic/immunologic, HEENT (head, ears, eyes, nose, throat), dermatologic/connective tissue, musculoskeletal, metabolic/nutritional, drug hypersensitivity, allergy, endocrine, major surgery, or other relevant diseases as revealed by history, physical examination, and laboratory assessments which may interfere with the absorption, distribution, metabolism or elimination of drugs or constituting a risk factor when taking the study medication
* A known history of epilepsy or with relatives with epilepsy
* Use of any drugs (prescribed and non-prescribed) within the last 2 weeks with the exception of paracetamol up to 48 hours before start of the study
* Any acute or chronic illness
* Participation in clinical trial or blood donation within 2 months before the study
* Drug and/or alcohol abuse or use of alcoholic beverages within 48 hours prior to the study or with a positive drug or alcohol test
* Use of tobacco or nicotine in any form or with a cotinine urinary level above 500 ng/ml
* Carriers of the Hepatitis B surface antigen (HBsAg) or carriers of the Hepatitis C or HIV virus
* A body temperature above 37.5 °C

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18
Dates: Start 2003-05; Study Completion 2003-11

PRIMARY OUTCOMES:
effect of SLV317 on substance P-induced venodilation

CONTACTS AND LOCATIONS:
Overall Officials: Walter E Haefeli, MD, Principal Investigator — Heidelberg University
Locations (1):
- Dept. of Internal Medicine VI, University of Heidelberg, Heidelberg, Baden-Wurttemberg, Germany